CLINICAL TRIAL: NCT05351463
Title: Papilla Suture Design Affects Papillary Postsurgical Dimensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Polak David, Principal Investigator, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-0079-15
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Periodontal Surgery; Oral Surgery

STUDY DESIGN:
Intervention Model Description: RCT parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm study (Other): in each case one site was assigned as control site and one site was assigned as test site.
  Interventions: Procedure: papila suture technique

INTERVENTIONS:
Procedure: papila suture technique — simple interupted vs internal horoizontal matress suture

SUMMARY:
The current prospective, randomized, controlled clinical trial aimed at comparing the impact of papillae suture technique on interdental papilla dimensions after periodontal surgery using a novel 3D intraoral scanning technique.

DETAILED DESCRIPTION:
Scientific rationale for study: Choosing the appropriate suture design for periodontal surgery may affect post-surgery tissue dimension. This is a critical issue in periodontal surgery due to the grave impact papilla play on soft tissue esthetics.

Principal findings: using the novel 3D scanning of the gingiva tissue show that simple interrupted suture negatively affect post-surgery papillary height and recession adjacent to the suture compared with vertical internal mattress suture.

Practical implications: the study provide evidence that allows the clinician to better choose the suture design that will allow optimal healing of the papilla. Furthermore, the study presents a novel 3D scanning method to analyzed dimensional changes in the soft tissue.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Systemically healthy (based on health questionnaire prior to treatment)
* Willingness to participate in the study
* Clinical requirement for periodontal\ implant surgery

Exclusion Criteria:

* Diagnosis of diabetes/heart disease, thrombocytopenia\ coagulation factors deficiency
* Chronic use\abuse of drugs\ alcohol
* Pregnancy Smoking more than 10 cigarettes per day Antibiotic consumption in the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
papilary volume | 12 weeks post surgery
  changes in papilary volume using 3D scanner

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No